CLINICAL TRIAL: NCT02505958
Title: How Quickly Can the Effects of Excessive Caloric Intake on Insulin Resistance be Reversed?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22331; R01DK090588 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: insulin resistance, obesity, caloric intake
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high caloric intake (Other): Volunteers will receive 3 meals and 3 snacks over a 24 hour period which will contain ~ 6,000 calories. Main meals will consist of ~ 1,500 calories and snacks will contain ~ 500 calories.
  Interventions: Other: high caloric intake
- reduced caloric intake (Other): On days 5 and 6 subjects will receive 3 meals only and each meal will contain ~ 333 calories for a total of 1,000/ 24 hours.
  Interventions: Other: reduced caloric intake

INTERVENTIONS:
Other: high caloric intake — Volunteers will be started on a diet program for 4 ½ days, consisting of 3 meals and 3 snacks over a 24 hour period and containing ~ 6000 Kcal/24 h.
  Arms: high caloric intake
Other: reduced caloric intake — On days 5 and 6, volunteers will received 3 meals (~333 calories each) totaling ~ 1,000 calories/24 hours.
  Arms: reduced caloric intake

SUMMARY:
Objective: To show that a 1-2 day reduction of caloric intake can reduce the insulin resistance produced by several days of overnutrition. Approach: Healthy volunteers will be admitted to the Clinical Research Center and undergo a baseline euglycemic-hyperinsulinemic clamp study to assess their insulin resistance. Subjects will then start on an overnutrition program for 4 days consisting of 3 meals and 3 snacks containing ~6,000 Kcal/24hours. A second clamp study will be performed on day 5 to demonstrate the overnutrition induced increase in insulin resistance. Starting on day 5 the subject's caloric intake will be reduced to ~1,000 Kcal for 2 days (day 5 and 6). After that on the morning of day 7, a third hyperinsulinemic-euglycemic clamp will be performed to determine whether the reduced caloric intake did reduce insulin resistance and the volunteer will be discharged from the Clinical Research Center.

DETAILED DESCRIPTION:
Study volunteers will be admitted to the Clinical Research Center at Temple University Hospital. After an overnight fast, body composition will be determined non-invasively by bioimpedance analysis (4) and a 4 h euglycemic-hyperinsulinemic clamp (using only FDA-approved regular insulin) as previously described (5) will be performed during which serum samples will be obtained for measurement of glucose, insulin, free fatty acids, ketone bodies and lipids. Oxidative stress ( 6) will be measured by 24 hour urine collections (analyzed for isoprostane content via 8-isoprostaglandin-F2alpha throughout the study period. Respiratory gas exchange rates (7) will be determined at hourly intervals (with a metabolic cart (True One, Parvo Utah) during the clamp studies and once a day on Days 2 through 6. After that, (at about 1:00 in the afternoon on Day 1) the volunteers will be started on a diet program for 4 ½ days, consisting of 3 meals and 3 snacks over a 24 hour period and containing ~ 6000 Kcal/24 h. The main meals (containing ~ 1500 Kcal/meal) will be served at ~ 8:00 in the morning (breakfast), 1:00 in the afternoon (lunch) and approximately 7:00 in the evening (dinner), the snacks (~ 500 Kcal/each) at approximately 11:00 in the morning, 4:00 in the afternoon and 11:00 in the night. On days 5 and 6, volunteers will receive 3 meals, each will contain ~333 calories. Each morning blood samples will be obtained to measure glucose insulin, free fatty acids and ketone bodies. Daily 24 h urine collections will be obtained each day. In the morning of Days 5 and 7, all procedures described for Day 1 will be repeated. In the afternoon of Day 7, the volunteers will be discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria: Healthy non-obese men and women -

Exclusion Criteria: Subjects with diabetes or a history of obesity surgery or with more than modest health problems

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin resistance | baseline, day 4 and day 7
  Insulin resistance will be determined by measuring changes in insulin-stimulated total body glucose uptake during euglycemic hyperinsulinemic clamping
Changes in oxidative stress | baseline, day1, day 2, day 3, day 4, day 5, day 6, day 7
  24 hour urine collections analyzed for isoprostane content
Changes in energy expenditure | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Changes in energy expenditure will be assessed with a metabolic cart (indirect calorimetry)
Changes in weight | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Subjects will be weighed daily
Changes in body composition | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Body composition will be determined by bioelectric impedance analysis

SECONDARY OUTCOMES:
Changes in blood glucose levels | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Daily blood samples will be analyzed to determine glucose levels of glucose.
Changes in blood levels of insulin | Baseline, day1 day2, day 3, day 4, day 5, day 6, day 7
  Daily blood samples will be analyzed to determine insulin levels
Changes in blood levels of free fatty acids | Baseline, day1 , day 2, day 3, day 4, day 5, day 6, day 7
  Daily blood samples will be analyzed to determine free fatty acid levels
Changes in blood ketone levels | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Daily blood samples will be analyzed to determine ketone levels
Changes in glucagon levels | baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Daily blood samples will be analyzed to determine glucagon levels

CONTACTS AND LOCATIONS:
Overall Officials: Ajaykumar Rao, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States